CLINICAL TRIAL: NCT07389720
Title: Characterization of (A)Typical Sensorimotor Pathways in Individuals With Autism
Acronym: MovAUT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 95/24 (ex 1105)
Record Dates: First submitted 2026-01-21; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; motor skills; social communication; kinematics
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Clinical, neuropsychological, neurophysiological, and genetic evaluations (Experimental): All children and their parents enrolled in the study will undergo an assessment of intellectual functioning, and a direct evaluation of motor skills using the Movement Assessment Battery for Children - Thirs Edition (MABC-3). Motor skills will also be assessed indirectly through either a parent or self-completed questionnaire. The motor profile of the participants will be further characterized using kinematic analysis of upper-limb movements during two experimental tasks.
  Interventions: Diagnostic Test: clinical assessment; Diagnostic Test: Neuropsychological examination; Diagnostic Test: Neurophysiological evaluation; Diagnostic Test: Genetic evaluation

INTERVENTIONS:
Diagnostic Test: clinical assessment — Clinical evaluation of participants by means of Autism Diagnostic Observation Schedule, Social Responsiveness Scale
Diagnostic Test: Neuropsychological examination — The participants' motor skills are measured using the Movement Assessment Battery for Children 3 (MABC3), the Developmental Coordination Disorder Questionnaire (DCDQ) or the Adult Developmental Coordination Disorder/Dyspraxia Checklist (ADC), and the kinematic analysis of upper-limb movements during two experimental tasks: (a) a reaching-and-inserting task involving a ball (ball task), and (b) a task requiring grasping a moving ball (ball-rolling task).
Diagnostic Test: Neurophysiological evaluation — Magnetic Resonance Imaging (structural MRI and spectroscopy)
Diagnostic Test: Genetic evaluation — Either blood or saliva will be obtained for participants for DNA collection. DNA will be extracted in the Molecular Biology Laboratory at the Scientific Institute IRCCS Medea. Captured exome libraries will be sequenced using the Illumina NextSeq 500 in 100 bp paired end reads. Postsequencing reads will be aligned using BWA Enrichment application on BaseSpace. Variant Call Format file will be then marked using wANNOVAR (Wang Genomics Lab). The analysis will be focused on non-synonymous variants enrichment in Gene Ontology and Human Phenotype

SUMMARY:
The goal of this interventional study is to understand whether sensorimotor skills could represent an endophenotype for autism, i.e. a specific class of biomarkers that bridges the gap between biological components of a condition and the behavioral/clinical dimensions. Motor and sensory differences are often observed in people with autism and may appear early in development or be shared among family members.

The study will address three main questions:

* What are the developmental effects of early differences in motor and sensory skills?
* Are motor and sensory abilities influenced by family relationships?
* Can studying motor and sensory differences in autism help researchers better understand the biological mechanisms underlying the condition? This study is structured in three topic-oriented work packages (WPs): WP1, a longitudinal assessment of sensorimotor skills as early predictors of later social characteristics in a mixed sample of infant siblings of autistic children (at elevated likelihood of autism) or with typical familial likelihood (no first-degree relatives with autism) (Q1); WP2, a cross-sectional investigation of sensorimotor abilities in autistic children and their parents as compared with typically developing children and their parents (Q2); and WP3, a dense-phenotyping approach to establish, within individuals, associations between traits across behavioral, neural, and molecular levels.

ELIGIBILITY:
Inclusion Criteria:

* children aged 2 to 12 years (both autistic and typically developing)
* Clinical diagnosis of Autism Spectrum Disorder based on clinical judgment according to DSM-5 criteria (for the autism group).
* being parents of the enrolled children (both autistic and typically developing)
* infants younger than 24 months of age with a first-degree family member with a clinical diagnosis of Autism Spectrum Disorder.

Exclusion Criteria:

* Presence of medical and/or neurological conditions of clinical significance, including epilepsy.
* Presence of dysmorphic syndromes or known genetic syndromes.
* Current use of medications and/or psychotropic drugs.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Movement Assessment Battery for Children 3 (MABC3) | immediately after the intervention
  The Movement ABC-3 (Movement Assessment Battery for Children, Third Edition) is a comprehensive, standardized assessment tool for identifying gross and fine motor coordination difficulties in individuals aged 3 to 25, assessing skills like dexterity, aiming, catching, balance, and locomotion.
Developmental Coordination Disorder Questionnaire (DCDQ) | immediately after the intervention
  The Developmental Coordination Disorder Questionnaire (DCDQ) is a parent questionnaire originally developed for estimating gross and fine motor skill difficulties in children. The questionnaire consists of 15 items investigating different subdomains of motor abilities, such as ball skills, complex motor coordination, fine and general motor skills. For each item, parents rate the children's degree of motor coordination on a 5-point scale comparing it to same-age peers.
Adult Developmental Coordination Disorder/Dyspraxia Checklist (ADC) | immediately after the intervention
  The Adult Developmental Coordination Disorder/Dyspraxia Checklist (ADC) is a self-report screening tool for adults (16+) to identify potential Developmental Coordination Disorder (DCD/Dyspraxia) by assessing lifelong motor challenges in daily activities
kinematic analysis of two motor tasks | immediately after the intervention
  (a) a reaching-and-inserting task involving a ball (ball task), which consists in reaching and grasping a rubber ball (diameter: 6 cm) placed over a support and dropping it in a small basket, provided with a hole large enough (diameter: 7 cm) not to require fine movements; (b) a task requiring grasping a moving ball (ball-rolling task) which requires participants to catch a ball rolling toward them on a curvilinear path off an inclined tabletop. As outcome measure, we will consider the total movement duration (recorded in sec).

SECONDARY OUTCOMES:
Magnetic Resonance (MRI) | immediately after the intervention
  Magnetic Resonance (MRI) of the Brain - MRI signal allowing tridimensional multiplanar reconstruction of the brain's structures. Anatomical images obtained with high definition T1 weighted sequences of radio frequencies - the measure is a "signal (in Hz) to noise ratio" which is obtained from each voxel (tiny 3D portions of the brain)
Magnetic Resonance Spectroscopy | immediately after the intervention
  Magnetic Resonance Spectroscopy (MRS) is a non-invasive technique, often used with MRI, that measures the chemical makeup (metabolites) of tissues like the brain.
Exome sequencing | immediately after the intervention
  Exome libraries will be sequenced using the Illumina NextSeq 500 in 100 bp paired end reads. Postsequencing reads will be aligned using BWA Enrichment application on BaseSpace. Variant Call Format file will be then marked using wANNOVAR (Wang Genomics Lab).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS E. Medea, Bosisio Parini, Lecco, Italy

IPD SHARING:
Plan to Share IPD: No